CLINICAL TRIAL: NCT02221154
Title: Use of Myo-inositol as Adjuvant Therapy in Patients With Polycystic Ovary Syndrome (PCOS) in Vitro Fertilization (IVF)
Acronym: FIV-INOPK
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHD 096-13
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2016-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: in vitro fertilization; ovarian hyperstimulation; pregnancy
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Gonadotropins; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inofolic® (Experimental): standard ovarian stimulation and Inofolic®
  Interventions: Dietary Supplement: Inofolic®; Other: Gonadotropins; Folic Acid
- Gonadotropins;Folic Acid (Active Comparator): standard ovarian stimulation without Inofolic®
  Interventions: Other: Gonadotropins; Folic Acid

INTERVENTIONS:
Dietary Supplement: Inofolic®
  Arms: Inofolic®
Other: Gonadotropins; Folic Acid — standard ovarian stimulation

SUMMARY:
The original mechanism of action of myo-inositol and preliminary results available in the literature on its use in IVF suggest its value as adjuvant gonadotropin therapy to reduce the risk of OHSS in PCOS patients.

The aim of the study is to demonstrate that administration of myo-inositol decreases the incidence of ovarian hyperstimulation syndrome (OHSS) in high-risk infertile with PCOS supported in IVF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients PCOS (Rotterdam ESHRE / ASRM criteria)

Combination of at least two of the following three criteria:

* Cycle disorder
* Clinical hyperandrogenism and / or biological
* Account antral follicles> 24
* Age ≤ 18 ≤ 38 years
* BMI <35 kg / m²
* Able to understand the protocol and signed informed consent

Exclusion Criteria:

* Patients not having the Rotterdam criteria
* Patients> 38 years and / or BMI> 35 kg / m²
* Woman enjoying a measure of legal protection
* Hypersensitivity to any component of the Inofolic (myo-inositol, soy, folic acid, glycerol, gelatin, coloring E171)
* Participation in another interventional biomedical research with treatment administered may disrupt ovarian stimulation

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-11; Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Incidence of OHSS in each group, graded mild, moderate or severe based on the recommendations | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne DELAY, PH, Principal Investigator — CHD Vendée La Roche sur Yon
Locations (4):
- France (4):
  - CHI de Créteil, Créteil
  - CHD Vendée, La Roche-sur-Yon
  - CHU de Nantes, Nantes
  - CH de Saint Nazaire, Saint-Nazaire